CLINICAL TRIAL: NCT05405712
Title: Increasing Peer Support for OUD Recovery During COVID-19 Through Digital Health: A National Randomized Controlled Trial
Brief Title: Mobile Peer Support for OUD Recovery
Acronym: MPS
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH); Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2105003009; R01DA054698-01 (NIH)
Record Dates: First submitted 2022-05-17; First posted 2022-06-06 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-10

CONDITIONS: Opioid Use Disorder
Keywords: drug overdose; substance-related disorders; chemically-induces disorders; Fentanyl; Analgesics, opioid; Narcotics; Naloxone; Central Nervous System Depressants; Physiological Effects of Drugs; Medications for Opioid Use Disorder; Recovery; Application; Machine-learning; Mobile treatment; Natural language processing; Opioid use disorder; Peer support; Technology
MeSH Terms: conditions — Opioid-Related Disorders; Drug Overdose; Substance-Related Disorders

STUDY DESIGN:
Intervention Model Description: Participants randomized to receive the APP intervention will receive login and sign up instructions to use the Marigold Health app. Both arms will receive standardized peer recovery support resources from SAMHSA
Who Masked: Investigator, Outcomes Assessor
Masking Description: The biostatistician will be blinded to the intervention/control group assignment throughout the course of the study and the assignments. Additionally, the principal investigator will remain blinded to the randomization.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Marigold APP (Experimental): Participants randomized to receive the APP will be enrolled in an app based peer support program
  Interventions: Behavioral: Mobile Phone App
- CONTROL (No Intervention): In the control arm participants will receive existing standardized peer recovery support resources from SAMHSA

INTERVENTIONS:
Behavioral: Mobile Phone App — App-based peer support program, used in conjunction with standard outpatient treatment
  Other Names: Peer Recovery App
  Arms: Marigold APP

SUMMARY:
The COVID-19 pandemic puts individuals recovering from opioid use disorders (OUDs), an already vulnerable population, at increased risk of overdose due to decreased access to treatment, decreased social support, and increased psychosocial stress. This proposal will test the efficacy of a promising mobile app-based peer support program, compared to usual care, in increasing recovery capital, improving retention in treatment, and reducing psychosocial adverse effects, among a national sample of people in recovery from OUD. If effective, it would provide an accessible, personalized, and scalable approach to OUD recovery increasingly needed during the COVID-19 pandemic.

DETAILED DESCRIPTION:
Increasing numbers of opioid overdoses have been observed during the COVID-19 pandemic, likely reflecting the pandemic's multiple effects on this already vulnerable population. People in recovery from opioid use disorder (OUD) have reported disproportionate psychosocial distress and isolation, as well as significant disruptions in access to treatment including peer support, during the COVID-19 pandemic. These negative outcomes are especially acute for rural, low-income, and minority populations in recovery from OUD. Peer support is a key component of many evidence-based OUD recovery programs: it improves recovery capital, improves treatment engagement, improves perceived social support, and reduces psychosocial distress, particularly when used in conjunction with other evidence-based treatments such as medication for opioid use disorder (MOUD). This grant, submitted in response to PA 20-237, therefore proposes a randomized controlled trial of a novel mobile peer support app platform among a national sample of 1300 patients in recovery from opioid use disorders (OUDs), as an adjunct to usual care, during COVID-19. The previously piloted online-only recruitment and follow-up strategy - in which investigators meld patient-reported outcomes with administrative datasets - allows strategic recruitment of often-excluded participants from across the United States, including those facing the highest barriers to treatment. The mobile app-based peer support intervention, provided as an individual-level enhancement of existing treatment and recovery programs, will allow individuals in OUD recovery to access a tailored, anonymous, peer-moderated support group 24/7. The app is augmented with natural language processing tools capable of automatically 'flagging' critical or clinically relevant content, thereby creating a scalable system to keep groups safe and constructive. Participants will be followed for 6 months through both self-report and administrative outcomes. The study's primary outcome is self-reported recovery capital, complemented by objectively measured administrative data on retention in treatment programs from our community and governmental partners in a sub-sample of 650 patients from RI and IN. Hypothesized secondary outcomes are mitigation of psychosocial effects of COVID-19 on this vulnerable population, including depressive symptoms, stress, and loneliness, as well as objective adverse events of emergency department visits and opioid overdoses. Finally, the investigators will explore whether state- and county-level variables moderate efficacy. OUD is a major public health problem, and patients in recovery from OUD are experiencing worse outcomes during the COVID-19 pandemic. If this mobile app demonstrates efficacy among a large national sample of patients, it has the potential to augment existing treatment programs, improve recovery capital, and reduce disproportionate impacts of COVID-19 on this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age ≥ 18 years old
* Own their own smartphone
* Self-identifying as being in recovery from or treatment for an opioid use disorder

Exclusion Criteria:

* Does not have an Android or iOS platform smartphone
* Previous enrollment in the study
* Currently incarcerated
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2022-05-12 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Change in the Brief Assessment of Recovery Capital (BARC-10) score over 6 month study period | 6 months
  This primary outcome measure will test the efficacy of app-based peer support, compared to the control, in improving recovery capital and engagement in treatment programs. The investigators will measure a change in the Brief Assessment of Recovery Capital (BARC-10) scores, between study groups over 6 months. The Brief Assessment of Recovery Capital will be asked at baseline, 1month follow up, 3 month follow up and 6 month follow up surveys. This score is an abbreviated 10-item measure of recovery capital with high internal consistency. The scale is from 1 "Strongly Disagree" to 6 "Strongly Agree." Total scores can range from 10 to 60. Scores of 47 or higher that are sustained over time indicate higher chances of long term recovery.

CONTACTS AND LOCATIONS:
Overall Officials: Megan Ranney, MD, MPH, Principal Investigator — Brown University
Locations (2):
- United States (2):
  - Indiana University, Indianapolis, Indiana
  - Brown University School of Public Health, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Scherzer CR, Ranney ML, Jain S, Bommaraju SP, Patena J, Langdon K, Nimaja E, Jennings E, Beaudoin FL. Mobile Peer-Support for Opioid Use Disorders: Refinement of an Innovative Machine Learning Tool. J Psychiatr Brain Sci. 2020;5(1):e200001. doi: 10.20900/jpbs.20200001. Epub 2020 Feb 3. PMID 32149192